CLINICAL TRIAL: NCT05198778
Title: An Open, Single Dose Designed Clinical Study to Evaluate Safety and Pharmacokinetic/Pharmacodynamic Characteristics After Oral Administration of URC102 in Patients With Renal Impairment Under Fasted Conditions and Healthy Adult Volunteers Under Fasted and Fed Conditions
Brief Title: A Safety, PK, PD and Food Effect Study of URC102 in Healthy Adults and Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JW21102
Record Dates: First submitted 2021-12-16; First posted 2022-01-20 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Healthy, Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — URC102

STUDY DESIGN:
Intervention Model Description: Parallel study between groups (crossover study within healthy patients)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1: Renal impairment patient (Experimental): Administer URC102, single-dose
  Interventions: Drug: URC102
- Test group 2: Renal impairment patient (Experimental): Administer URC102, single-dose
  Interventions: Drug: URC102
- Control group: Healthy adult people (Experimental): Administer URC102, 2 doses
  Interventions: Drug: URC102

INTERVENTIONS:
Drug: URC102 — tablet
Drug: URC102 — tablet
  Arms: Control group: Healthy adult people

SUMMARY:
A phase 1 clinical trial to evaluate safety, PK/PD profiles and food effects of URC102 in patients with renal impairment and healthy people.

DETAILED DESCRIPTION:
This trial will evaluate

1. in patients with renal impairment: the safety, pharmacokinetics and pharmacodynamics after single oral administration of URC102 under fasted conditions.
2. in healthy adult subjects: the safety, pharmacokinetics and pharmacodynamics of 2 single doses of URC102 in the morning after fasting or after a high-fat breakfast. The 2 doses will be separated by a washout period.

ELIGIBILITY:
Inclusion Criteria:

For Test Group 1 and 2 - subjects with renal impairment

1. Age 19~65
2. BMI 18.0~30.0 kg/m^2 (Body mass index)
3. 30 ≤ eGFR < 60 mL/min/1.73m^2 (estimated glomerular filtration rate)
4. voluntarily given written informed consent

For Control Group - healthy subjects

1. Age ≥ 19
2. BMI 18.0~30.0 kg/m^2
3. eGFR ≥ 90 mL/min/1.73m^2
4. voluntarily given written informed consent

Exclusion Criteria:

For Test Group 1 and 2 - subjects with renal impairment

1. Medical history

   * Subjects with lactic acidosis or marked hepatotoxicity
   * Not controlled diabetes, hypertension, dyslipidemia
   * requiring dialysis
2. Clinical examination

   * AST, ALT > 2, Bilirubin total, γ-GTP > 1.5, CK > 2 times the upper limit of normal ranges (Aspartate transaminase, Alanine transaminase, gamma-Glutamyl transpeptidase, Creatine phosphokinase)
   * Positive serologic results
3. Drug hypersensitivity and drug abuse

For Control Group - healthy subjects

1. Medical history

   * History of chronic liver disease, hepatic encephalopathy, ascites, or upper gastrointestinal bleeding
   * Subjects with lactic acidosis or marked hepatotoxicity
2. Clinical examination

   * AST, ALT > 2, Bilirubin total, γ-GTP > 1.5, CK > 2 times the upper limit of normal ranges
   * Positive serologic results
3. Drug hypersensitivity and drug abuse

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from the point of administration to last time point of blood sampling (AUC) of UR-1102 | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48, 72 hours
  Pharmacokinetic parameter
Maximum concentration of drug in plasma (Cmax) of UR-1102 | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48, 72 hours
  Pharmacokinetic parameter

SECONDARY OUTCOMES:
Serum uric acid | 0, 2, 4, 6, 8, 10, 24, 48, 72 hours
  Pharmacodynamic parameter
Excretion amount of uric acid | 0, 2, 4, 6, 8, 10, 24, 48, 72 hours
  Pharmacodynamic parameter
Number of participants with treatment-related adverse events | up to 2 weeks
  Safety variable
Number of participants with clinical significant results of Physical examination | up to 2 weeks
  Safety variable
Number of participants with clinical significant results of Vital signs | up to 2 weeks
  Safety variable
Number of participants with clinical significant results of Laboratory tests | up to 2 weeks
  Safety variable

CONTACTS AND LOCATIONS:
Overall Officials: Min-kyu Park, MD, Principal Investigator — Chungbuk National University Hospital
Locations (2):
- South Korea (2):
  - Chungbuk National University Hospital, Cheongju-si
  - Ajou University Hospital, Suwon